CLINICAL TRIAL: NCT03299335
Title: Molecular Profile of the Evolution of Inclusion Body Myositis
Acronym: IBM-RNAseq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOI-05
Record Dates: First submitted 2017-09-20; First posted 2017-10-03 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early-stage sIMB patients (Other)
  Interventions: Other: Blood collection
- Late-stage sIMB patients (Other)
  Interventions: Other: Blood collection
- Control subjects (Other)
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — assay of CPK and anti-cN-1A antibodies

SUMMARY:
This study aims at assessing the gene expression in the muscles of patients suffering from sporadic Inclusion Body Myositis (sIBM) at various stages of the disease, by comparison with muscles of control subject. The investigators use the RNA-seq technique to analyze the gene expression levels and potential alternate transcripts, including long non-coding RNAs (lncRNAs), in muscle tissue samples. The gene expression profiles will point to the genes of interest that can then become the object of future studies, in which epigenetic changes of these genes will be explored further. The value of those possible biomarkers will be assessed. The investigators will also evaluate the correlation between the gene expression profile, the degree of functional impairment, the histological picture and the presence or absence of autoantibodies.

DETAILED DESCRIPTION:
Sporadic inclusion body myositis (sIBM) is a myopathy that usually does not become apparent before the age of 50 to 60. The disease is characterized by a progressive weakening of the muscles, including the finger flexors of the hand and proximal leg muscles. Swallowing problems are often observed. Muscular biopsy also reveals a combination of inflammatory, mitochondrial and myodegenerative signs. What triggers the disease has not yet been established, although two hypotheses are currently being explored: auto-immune and degeneration etiologies. Histological inflammatory hallmarks, the presence of sIMB-specific antibodies and the concomitance of other autoimmune pathologies point to the autoimmune hypothesis. On the other hand, immunosuppressive drugs only have a positive effect in a limited number of cases. The degenerative hypothesis is supported by the presence of rimmed vacuoles and protein aggregates (inclusion bodies) in the myocytes. The presence of mitochondrial anomalies can enhance protein aggregation that in turn can worsen mitochondrial changes.

Many genetic studies have been carried out to assess a potential genetic link in the sIBM. However, only connections to a number of HLA alleles and haplotypes have been found. In the present study, the investigators propose to evaluate gene expression in the muscular tissue by high-throughput RNA-sequencing (RNA-seq) in order to increase our knowledge of the sIMB pathophysiology. The RNA-seq technique can not only identify transcripted genes in a given tissue, but also discover unreported alternate or new transcripts, including long non-coding RNAs (lncRNAs). Indeed, lncRNAs play an important role in regulating gene networks, in particular in contributing to the setup and maintenance of epigenetic marks. The RNAseq approach will allow the investigators to assess the perturbations in the gene expression profiles and lncRNAs involved in the onset of the disease, by comparing the profiles obtained from patients at various stages of the disease and control subjects.

This study aims at assessing the gene expression in the muscles of patients suffering from sporadic Inclusion Body Myositis (sIBM) at various stages of the disease, by comparison with muscles of control subject. The investigators use the RNA-seq technique to analyze the gene expression levels and potential alternate transcripts, including long non-coding RNAs (lncRNAs), in muscle tissue samples. The gene expression profiles will point to the genes of interest that can then become the object of future studies, in which epigenetic changes of these genes will be explored further. The value of those possible biomarkers will be assessed. The investigators will also evaluate the correlation between the gene expression profile, the degree of functional impairment, the histological picture and the presence or absence of autoantibodies.

The study is interventional with no immediate benefits to the patient. RNAseq will be performed in both a group of sIBM patients (at early and late stages) and a group of control subjects.

Patients suffering from sIMB will be recruited on the basis of the ENMC 2011 diagnostic criteria. Predominant inflammatory changes (T-cell inflammatory infiltrate, expression of HLA class I antigens) without a degenerative affection (rimmed vacuoles, endomysial fibrosis, protein accumulation) will allow for a classification in the "early sIMB" group. Muscle biopsies of control subjects are part of a proprietary collection of the Neurology Department declared to the Nice University Hospital administration; they are selected from biopsies devoid of anomalies among subjects matching the ages of the sIMB patients. A physical examination and a venipuncture will be performed on patients in order to assess the absence or presence of anti-cN-1A antibodies, a new marker of sIMB. Control subjects will undergo a physical exam and a creatine kinase dosage. Tissue muscle has been collected beforehand in the frame of the routine diagnostic procedure for both patients and control subjects.

Expression profiles will be obtained by RNAseq from 15 muscle biopsies. Three groups of samples will be compared: 5 from early-stage sIMB patients, 5 from late-stage sIMB patients and 5 from control subjects.

In addition to known expression modifications of genes involved in the inflammatory response, in particular at early stages of the sIMB, or of genes involved in autophagy processes, at late stages of the disease where muscle degeneration is advanced, this study will allow identifying lncRNA potentially involved in the sIMB. Inasmuch as lncRNA are crucial for the regulation of cell differentiation and ageing processes at the epigenetic level, this pilot study will make possible to identify a group of genes of particular relevance, thus enabling further research on epigenetic regulation. Furthermore, a delayed gene expression, as is the case with lncRNA in early-stage sIMB patients, compared to lncRNA in late-stages disease patients, may prove a biomarker for evolution, and serve as a beneficial tool for monitoring sIMB in therapeutic trials to come.

ELIGIBILITY:
Inclusion Criteria (early-stage sIBM patients):

* Patient suffering from sIMB according to the ENMC 2011 criteria: "sIMB defined on histological and clinical features" with, on the inclusion visit day:

  * duration of the disease > 12 months;
  * onset of the disease > 45 years;
  * quadriceps weakness ≥ hip flexors and/or fingers flexors weakness > shoulder abductors;
  * CPK ≤ 15 x ULN.
* Patient with available biopsy showing alterations compatible with an inflammatory myopathy (endomysial inflammatory infiltrate, overexpression of HLA class I), but not specific to sIMB, in particular with no associated degenerative and/or mitochondrial pathologies (protein aggregates: amyloid, p62, SMI-31, TDP-43; 15-18nm filaments; ragged red fibers; COX negative fibers).
* Patient whose sIMB diagnosis has been histologically confirmed with a second muscle biopsy showing the typical histological hallmarks (endomysial inflammatory infiltrate, overexpression of HLA class I and an associated degenerative and/or mitochondrial pathology).
* Patient who gave his consent for the use of the biological material from the muscle biopsy at the time of the diagnosis.
* Patient affiliated to a social security regimen.
* Signed and written informed consent.

Exclusion Criteria (early-stage sIBM patients):

* Patient with a known medical record that could significantly influence the results of the study: auto-immune disease with conjunctive tissue inflammation (overlap myositis, rheumatoid arthritis, lupus, vasculitis, spondylarthritis, scleroderma, psoriatic arthritis), disease causing nerve-damage (Parkinson's disease, Alzheimer's disease, amyotrophic lateral sclerosis), auto-immune neuropathy (chronic polyradiculoneuritis and variants (multifocal motor neuropathy with conduction blocks, anti-MAG neuropathy)).
* Presence of the following histological characteristics in the muscle biopsy pointing to degenerative and/or mitochondrial pathologies: protein aggregates (amyloid, p62, SM-31, TDP-43), 15-18nm filaments, ragged red fibers or fibers with decreased COX activity.
* Patient who received one of the following treatments, prior to the first muscle biopsy:

  * anti-inflammatory drugs in the past week;
  * corticotherapy in the past month;
  * immunosuppressive agents in the past 3 months;
  * other treatments: chloridin, amiodarone, colchicine, vincristine in the past 6 months.
* Patient under curators or guardianship.
* Pregnant woman.

Inclusion Criteria (late-stage sIMB patients):

* Patient suffering from sIMB according to the ENMC 2011 criteria: "sIMB defined on histological and clinical features" with, on the inclusion visit day:

  * duration of the disease > 12 months;
  * onset of the disease > 45 years;
  * quadriceps weakness ≥ hip flexors and/or fingers flexors weakness > shoulder abductors;
  * CPK ≤ 15 x ULN.
* Patient whose sIMB diagnosis has been histologically confirmed with a muscle biopsy featuring the following characteristics: endomysial inflammatory infiltrate, rimmed vacuoles and protein aggregates (amyloid, p62, SM-31, TDP-43) or presence of 15-18nm filaments.
* Patient who gave his consent for the use of the biological material from the muscle biopsy at the time of the diagnosis.
* Patient affiliated to a social security regimen.
* Signed and written informed consent.

Non-inclusion criteria (late-stage sIMB patients):

* Patient with a known medical record that could significantly influence the results of the study: auto-immune disease with conjunctive tissue inflammation (overlap myositis, rheumatoid arthritis, lupus, vasculitis, spondylarthritis, scleroderma, psoriatic arthritis), disease causing nerve-damage (Parkinson's disease, Alzheimer's disease, amyotrophic lateral sclerosis), auto-immune neuropathy (chronic polyradiculoneuritis and variants (multifocal motor neuropathy with conduction blocks, anti-MAG neuropathy)).
* Patient who received one of the following treatments, prior to the muscle biopsy that confirmed the diagnosis:

  * anti-inflammatory drugs in the past week;
  * corticotherapy in the past month;
  * immunosuppressive agents in the past 3 months;
  * other treatments: chloridin, amiodarone, colchicine, vincristine in the past 6 months.
* Patient under curators or guardianship.
* Pregnant woman.

Inclusion Criteria (control subjects):

* Signed and written informed consent for the use of muscle tissue used collected for the diagnosis of a CPK elevation and/or myopathy and/or myalgias.
* No signs of muscular weakness at the time of the muscle biopsy.
* Age > 45, correlated to the age of sIMB patients, allowing for the constitution of a homogeneous group compared to sIMB patients.
* Patient affiliated to a social security regimen.
* Signed and written informed consent.

Non-inclusion criteria (control subjects):

* Subject with a muscle biopsy showing signs of inflammation and/or vacuoles and/or dystrophy.
* Subject with a known medical record that could significantly influence the results of the study: auto-immune disease with conjunctive tissue inflammation (overlap myositis, rheumatoid arthritis, lupus, vasculitis, spondylarthritis, scleroderma, psoriatic arthritis), disease causing nerve-damage (Parkinson's disease, Alzheimer's disease, amyotrophic lateral sclerosis), auto-immune neuropathy (chronic polyradiculoneuritis and variants (multifocal motor neuropathy with conduction blocks, anti-MAG neuropathy)).
* Subject with a confirmed sIMB diagnosis.
* Patient who received one of the following treatments, prior to the muscle biopsy that confirmed the diagnosis:

  * anti-inflammatory drugs in the past week;
  * corticotherapy in the past month;
  * immunosuppressive agents in the past 3 months;
  * other treatments: chloridin, amiodarone, colchicine, vincristine in the past 6 months.
* Patient under curators or guardianship.
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
sIBM gene expression profile | at 12 Months
  The expression of different genes in muscle tissue will be evaluated by RNA-seq and will allow to establish the IBM gene expression profile

SECONDARY OUTCOMES:
CPK level | at 12 Months
  The CPK level will be evaluated.
Rate of cN-1A antibodies. | at 12 Months
  Presence or absence of cN-1A antibodies will be evaluated.
IWCI score | at 12 Months
  The IWCI score will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pasteur 2 - Service Système Nerveux Périphérique, Muscle et SLA, Nice, France